CLINICAL TRIAL: NCT06667063
Title: Clinical Study on the Immune Response Characteristics of Novel Coronavirus and Influenza Virus Infection
Status: Recruiting | Type: Observational
Sponsor: Zhongnan Hospital (Other)
Collaborators: Institute of Biotechnology, Academy of Military Medical Sciences, PLA of China (Other)
Responsible Party: Principal Investigator, Jianying Huang, Chief Physician, Zhongnan Hospital
Other Study IDs: AMMS85-2401
Record Dates: First submitted 2024-10-07; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: COVID-19; Influenza
Keywords: COVID-19; Influenza; Immune response characteristics; Clinical study
MeSH Terms: conditions — COVID-19; Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples With DNA — Nasal mucosa/Nasopharyngeal mucosa/Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Cohort 1:COVID-19 infected persons: Inclusion Criteria:
  1. volunteers aged 18 years and above at the time of screening;
  2. informed consent obtained from volunteers and volunteers/witnesses able to sign the informed consent form;
  3. an interval of ≥3 months from the last COVID-19 or influenza vaccination;
  4. an interval of ≥ 3 months from the last respiratory viral infection such as COVID-19 or Influenza virus occurs;
  5. COVID-19 antigen-positive and within 48 hours of onset of symptoms of infection;
  Interventions: Other: Nasal swab/Nasopharyngeal swab/Blood sample collection
- Cohort 2:Influenza virus infected persons: Inclusion Criteria:
  1. volunteers aged 18 years and above at the time of screening;
  2. informed consent obtained from volunteers and volunteers/witnesses able to sign the informed consent form;
  3. an interval of ≥3 months from the last COVID-19 or influenza vaccination;
  4. an interval of ≥ 3 months from the last respiratory viral infection such as COVID-19 or Influenza virus occurs;
  5. influenza virus antigen-positive and within 48 hours of onset of symptoms of infection;
  Interventions: Other: Nasal swab/Nasopharyngeal swab/Blood draw
- Cohort 3:Healthy Volunteers: Inclusion Criteria:
  1. volunteers aged 18 years and above at the time of screening;
  2. informed consent obtained from volunteers and volunteers/witnesses able to sign the informed consent form;
  3. an interval of ≥3 months from the last COVID-19 or influenza vaccination;
  4. an interval of ≥ 3 months from the last respiratory viral infection such as COVID-19 or Influenza virus occurs;
  5. COVID-19 and influenza virus antigen-negative, no febrile symptoms, and no symptoms of viral or bacterial respiratory infections.
  Interventions: Other: Nasal swab/Nasopharyngeal swab/Blood draw

INTERVENTIONS:
Other: Nasal swab/Nasopharyngeal swab/Blood sample collection — Collect nasal or nasopharyngeal swab samples, 15ml anticoagulant samples and 3ml procoagulant samples, as well as 2ml blood samples for blood routine testing and C-reactive protein testing
  Groups: Cohort 1:COVID-19 infected persons
Other: Nasal swab/Nasopharyngeal swab/Blood draw — Visit 1/2/3：Collect nasal or nasopharyngeal swab samples, 15ml anticoagulant samples and 3ml procoagulant samples, as well as 2ml blood samples for blood routine testing and C-reactive protein testing
  Groups: Cohort 2:Influenza virus infected persons
Other: Nasal swab/Nasopharyngeal swab/Blood draw — Visit 1/2/3：Collect nasal or nasopharyngeal swab samples, 15ml anticoagulant samples and 3ml procoagulant samples, as well as 2ml blood samples for blood routine testing and C-reactive protein testing
  Groups: Cohort 3:Healthy Volunteers

SUMMARY:
This is an open-label, prospective observational study in people 18 years of age and older designed to track changes in the dynamics of the respiratory and peripheral blood immune response in people infected with influenza virus and new coronaviruses, and to resolve the characteristics of the virus-induced natural immune response.

DETAILED DESCRIPTION:
The clinical trial enrolls 130 subjects aged 18 years and older with ≥3 months between their last COVID-19/influenza vaccination or respiratory virus infection. Mucosal and peripheral blood samples will be collected from COVID-19-infected and influenza-infected patients during the preinfection, infection, and recovery periods, and cytokines, immune cell typing, immune cell transcription, and specific antibody levels will be examined in these patients. Levels of cytokines, immune cell typing, immune cell gene transcription, specific antibodies, etc.

ELIGIBILITY:
Inclusion Criteria:

1. volunteers aged 18 years and above at the time of screening;
2. informed consent obtained from volunteers and volunteers/witnesses able to sign the informed consent form;
3. an interval of ≥3 months from the last COVID-19 or influenza vaccination;
4. an interval of ≥ 3 months from the last respiratory viral infection such as COVID-19 or Influenza virus occurs; 5.1 cohort 1：novel coronavirus virus antigen-positive and within 48 hours of onset of symptoms of infection; 5.2 cohort 2：influenza virus antigen-positive and within 48 hours of onset of symptoms of infection; 5.3 cohort 3：novel coronavirus and influenza virus antigen-negative, no febrile symptoms, and no symptoms of viral or bacterial respiratory infections.

Exclusion Criteria:

1. known or suspected concomitant more serious and medically unstable disease in the judgment of the investigator, including: respiratory disease, tuberculosis, acute infections or active chronic disease, hepatic or renal disease, cardiovascular disease (cardiorespiratory failure), hypertension (systolic blood pressure ≥160 mmHg, diastolic blood pressure ≥100 mmHg), malignant tumors, infectious or allergic skin diseases, and the presence of HIV infection;
2. Absence of spleen or functional absence of spleen;
3. immunosuppressive therapy, anti-allergy therapy, cytotoxic therapy, inhaled corticosteroids (excluding corticosteroid spray therapy for allergic rhinitis, and superficial corticosteroid therapy for acute uncomplicated dermatitis) within the past 6 months;
4. Received blood products within the past 3 months;
5. has received other vaccines or investigational drugs within the past 1 month;
6. is receiving anti-tuberculosis treatment;
7. In the judgment of the investigator, due to a variety of medical, psychological, social, or other conditions that are contrary to the trial protocol or that affect the signing of informed consent by the volunteer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study is planned to include 50 patients infected with novel coronavirus, 50 patients infected with influenza virus and 30 healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The frequency of DC, monocyte, NK cell, macrophage cell, B cell and T cell in mucosal sample as calculated by Illumina NGS platform. | From the enrollment to the end of the visit on the 28th ± 3rd day
  Measuring method: Single-cell RNA sequencing. Metric/method of measurement: cell frequency
The Ct value of SARS-CoV-2 N gene, Influenza A HA gene and Influenza B PA gene in mucosal sample as assessed by Real-Time RT-PCR | From the enrollment to the end of the visit on the 28th ± 3rd day
  Measuring method: Real-Time RT-PCR Metric/method of measurement: Ct value
The SARS-CoV-2, Influenza A and Influenza B-specific IgG titer in serum sample assessed by ELISA. | From the enrollment to the end of the visit on the 28th ± 3rd day
  Measuring method: ELISA Metric/method of measurement: antibody titer
The level of IL-1β, IL-6, IFN-gamma, MCP-1, CXCL9, CXCL10, MCP-1 and TNF-alpha in serum sample assessed by Luminex. | From the enrollment to the end of the visit on the 28th ± 3rd day
  Measuring method: Luminex Metric/method of measurement: concentration
The transcriptome profiles of peripheral blood mononuclear cell assessed by RNA-sequencing Measuring method: RNA-sequencing | From the enrollment to the end of the visit on the 28th ± 3rd day
  Metric/method of measurement: gene count
The frequency of DC, monocyte, NK cell, macrophage cell, B cell and T cell in blood sample as assessed by the flow cytometer | From the enrollment to the end of the visit on the 28th ± 3rd day
  Measuring method: flow cytometer Metric/method of measurement: cell frequency

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wimmers F, Donato M, Kuo A, Ashuach T, Gupta S, Li C, Dvorak M, Foecke MH, Chang SE, Hagan T, De Jong SE, Maecker HT, van der Most R, Cheung P, Cortese M, Bosinger SE, Davis M, Rouphael N, Subramaniam S, Yosef N, Utz PJ, Khatri P, Pulendran B. The single-cell epigenomic and transcriptional landscape of immunity to influenza vaccination. Cell. 2021 Jul 22;184(15):3915-3935.e21. doi: 10.1016/j.cell.2021.05.039. Epub 2021 Jun 25. PMID 34174187
- [Background] Su Y, Chen D, Yuan D, Lausted C, Choi J, Dai CL, Voillet V, Duvvuri VR, Scherler K, Troisch P, Baloni P, Qin G, Smith B, Kornilov SA, Rostomily C, Xu A, Li J, Dong S, Rothchild A, Zhou J, Murray K, Edmark R, Hong S, Heath JE, Earls J, Zhang R, Xie J, Li S, Roper R, Jones L, Zhou Y, Rowen L, Liu R, Mackay S, O'Mahony DS, Dale CR, Wallick JA, Algren HA, Zager MA; ISB-Swedish COVID19 Biobanking Unit; Wei W, Price ND, Huang S, Subramanian N, Wang K, Magis AT, Hadlock JJ, Hood L, Aderem A, Bluestone JA, Lanier LL, Greenberg PD, Gottardo R, Davis MM, Goldman JD, Heath JR. Multi-Omics Resolves a Sharp Disease-State Shift between Mild and Moderate COVID-19. Cell. 2020 Dec 10;183(6):1479-1495.e20. doi: 10.1016/j.cell.2020.10.037. Epub 2020 Oct 28. PMID 33171100
- [Background] Clementi N, Ghosh S, De Santis M, Castelli M, Criscuolo E, Zanoni I, Clementi M, Mancini N. Viral Respiratory Pathogens and Lung Injury. Clin Microbiol Rev. 2021 Mar 31;34(3):e00103-20. doi: 10.1128/CMR.00103-20. Print 2021 Jun 16. PMID 33789928